CLINICAL TRIAL: NCT01264354
Title: An Open Study to Evaluate the Efficacy, Safety of Clevudine Monotherapy or Adefovir and Clevudine Combination in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Byung Chul Yoo/Samsung Medical Center, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLV-412
Record Dates: First submitted 2010-12-19; First posted 2010-12-21 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — clevudine; adefovir dipivoxil; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Clevudine 30mg
  Interventions: Drug: Clevudine 30mg
- 2 (Experimental): Clevudine 20mg+Adefovir dipivoxil 10mg
  Interventions: Drug: Clevudine 20mg+Adefovir dipivoxil 10mg
- 3 (Experimental): Clevudine 20mg
  Interventions: Drug: Clevudine 20mg

INTERVENTIONS:
Drug: Clevudine 30mg — Clevudine 30mg
  Other Names: Levovir 30mg
  Arms: 1
Drug: Clevudine 20mg+Adefovir dipivoxil 10mg — Clevudine 20mg+ Adefovir 10mg
  Other Names: Levovir 20mg+Adefovir 10mg
  Arms: 2
Drug: Clevudine 20mg — Clevudine 20mg
  Other Names: Levovir 20mg
  Arms: 3

SUMMARY:
This is an open study to evaluate the efficacy, safety of clevudine monotherapy or adefovir and clevudine combination in patients with chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years and older.
* Patient is documented to be HBsAg positive for > 6 months.
* Patient is HBV DNA positive with DNA levels ≥ 1×10^5 copies/mL within 30days of baseline.
* Patient has ALT levels ≥ 1×ULN
* Patient who is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

* Patient is currently receiving antiviral, immunomodulatory, cytotoxic or corticosteroid therapy.
* Patients previously treated with interferon, peg-interferon or other immunomodulatory within the previous 6 months.
* Patients previously treated with clevudine, lamivudine, adefovir, entecavir, telbivudine, Tenofovir or any other investigational nucleoside for HBV infection.
* Patient with clinical evidence of decompensated liver disease (Total bilirubin < 2.0mg/dL, Prothrombin time < 1.7(INR), Serum albumin≥3.5g/dL)
* Patient is coinfected with HCV, HDV or HIV.
* Patient has a history of ascites, variceal hemorrhage or hepatic encephalopathy.
* Patient with clinical evidence of hepatocellular carcinoma
* Patient with previous liver transplantation
* Patient is pregnant or breast-feeding.
* Patient has a clinically relevant history of abuse of alcohol or drugs.
* Patient has a significant immunocompromised, gastrointestinal, renal,
* hematological, psychiatric, bronchopulmonary, biliary diseases excluding asymptomatic GB stone, neurological, cardiac, oncologic(except HCC)or allergic disease or medical illness that in the investigator's opinion might interfere with therapy.
* Patient has creatinine clearance less than 60mL/min as estimated by the following formula: (140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-08 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HBV DNA levels < 300 copies/mL | 24 week

SECONDARY OUTCOMES:
The change of HBV DNA form the baseline | 24week, 48week, 96week
  (log copies/mL)
Proportion of patients with HBV DNA < 300 copies/mL | 48week, 96week
Proportion of patients with ALT normalization | 24week, 48week, 96week
Proportion of patients with HBeAg loss and/or seroconversion | 96 Week

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea